CLINICAL TRIAL: NCT07315217
Title: Cortical Excitability and Role of Non Invasive Brain Stimulation in ADHD and AUTISM : Double Blind Randomized Clinical Trial
Brief Title: Cortical Excitability and Role of Non Invasive Brain Stimulation in ADHD and AUTISM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amaal Emad Khairy, Resident at Neuropsychiatry Department, Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Brain Stimulation in ADHD/ASD
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Cortical Excitability; Brain Stimulation; ADHD; Autism
Keywords: Cortical excitability; non invasive brain stimulation; ADHD; Autism
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Autistic Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ADHD Active rTMS (Experimental): Children and adolescents with ADHD receive high-frequency rTMS over the right dorsolateral prefrontal cortex (10 Hz, 1200-1500 pulses per session, 100-110% of resting motor threshold) for 15 sessions over 3 weeks in addition to standard care.
  Interventions: Device: Active repetitive transcranial magnetic stimulation (rTMS)
- ADHD Sham rTMS (Sham Comparator): Children and adolescents with ADHD receive sham rTMS using the same session schedule and procedures as the active ADHD rTMS arm, with coil positioning and sound mimicking stimulation but without effective magnetic pulses, plus standard care.
  Interventions: Device: Sham repetitive transcranial magnetic stimulation (sham rTMS)
- ASD Active rTMS (Experimental): Children and adolescents with autism spectrum disorder receive low-frequency (1 Hz) or intermittent theta-burst rTMS over bilateral dorsolateral prefrontal cortex (about 1200 pulses per session) for 15 sessions over 3 weeks, according to the protocol and ethical approval, plus standard care.
  Interventions: Device: Active repetitive transcranial magnetic stimulation (rTMS)
- ASD Sham rTMS (Sham Comparator): Children and adolescents with autism spectrum disorder receive sham rTMS over bilateral dorsolateral prefrontal cortex with identical session number and duration as the active ASD rTMS arm, but without effective stimulation, plus standard care.
  Interventions: Device: Sham repetitive transcranial magnetic stimulation (sham rTMS)

INTERVENTIONS:
Device: Active repetitive transcranial magnetic stimulation (rTMS) — Active repetitive transcranial magnetic stimulation delivered using a figure-of-eight coil. For ADHD, high-frequency 10 Hz rTMS is applied over the right dorsolateral prefrontal cortex at 100-110% resting motor threshold, 1200-1500 pulses per session, 15 sessions over 3 weeks. For ASD, 1 Hz inhibitory rTMS or intermittent theta-burst stimulation is applied over bilateral dorsolateral prefrontal cortex with approximately 1200 pulses per session, 15 sessions over 3 weeks.
  Arms: ADHD Active rTMS; ASD Active rTMS
Device: Sham repetitive transcranial magnetic stimulation (sham rTMS) — Sham rTMS using the same device and schedule as active treatment, with coil positioning and acoustic cues mimicking stimulation but without delivering effective magnetic pulses. Fifteen sham sessions are administered over 3 weeks for ADHD and ASD participants in the sham arms, in addition to standard clinical care.
  Arms: ADHD Sham rTMS; ASD Sham rTMS

SUMMARY:
This double-blind, randomized, sham-controlled clinical trial will evaluate the effects of repetitive transcranial magnetic stimulation (rTMS) on children and adolescents with attention-deficit/hyperactivity disorder (ADHD) or autism spectrum disorder (ASD) and matched healthy controls. Participants aged 6-19 years will be assigned to active or sham rTMS protocols targeting the dorsolateral prefrontal cortex over 3 weeks, with assessment of changes in disorder-specific symptoms and cortical excitability. The study aims to determine the safety, feasibility, and preliminary efficacy of rTMS as a non-invasive neuromodulation approach in pediatric neurodevelopmental disorders.

DETAILED DESCRIPTION:
Altered cortical excitability and imbalance between excitation and inhibition have been reported in both ADHD and ASD, suggesting that non-invasive brain stimulation may modulate underlying pathophysiology. This study comprises two parallel, double-blind, sham-controlled rTMS trials in children and adolescents aged 6-19 years with ADHD or ASD and age- and sex-matched healthy controls. In the ADHD cohort, high-frequency 10 Hz rTMS will be delivered over the right dorsolateral prefrontal cortex, whereas in the ASD cohort low-frequency 1 Hz or intermittent theta-burst rTMS will be delivered over bilateral dorsolateral prefrontal cortex, each for 15 sessions over 3 weeks. Sham stimulation will mimic sound and procedure without effective magnetic pulses.

Cortical excitability will be assessed using single- and paired-pulse TMS measures (such as resting motor threshold, short-interval intracortical inhibition, long-interval intracortical inhibition, cortical silent period, and transcallosal inhibition). Blood samples will be collected to measure dopamine and brain-derived neurotrophic factor as potential neurochemical correlates. Primary clinical outcomes are changes in validated ADHD and ASD symptom rating scales, with secondary outcomes including changes in cortical excitability indices, biomarker levels, and safety/tolerability events. Data will be collected in a secure database and analyzed with mixed-effects models to estimate treatment effects and generate effect-size estimates to inform future definitive trials of rTMS in pediatric neurodevelopmental disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-19 years.
* ASD trial: DSM-5 diagnosis of ASD confirmed by CARS-2.
* ADHD trial: DSM-5 diagnosis of ADHD confirmed by structured interview/CONORS
* IQ ≥ 70.
* Stable medication for ≥4 weeks (if any).

Exclusion Criteria:

* Epilepsy or seizure history.
* Metallic implants or devices incompatible with TMS.
* Severe psychiatric comorbidity (e.g., psychosis).
* Inability to tolerate TMS procedures.

Ages: 6 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change in ADHD symptom severity | Baseline (pre-treatment) and within 1 week after completion of the 3-week rTMS/sham treatment course.
  Mean change in total score on a validated ADHD rating scale (for example, Conners' Parent Rating Scale) from baseline to end of treatment, comparing active rTMS with sham in children and adolescents with ADHD. The primary analysis will use mixed-effects models including fixed effects for group (active vs sham), time, and group × time interaction to estimate the treatment effect on ADHD symptom severity.
Change in autism symptom severity | Baseline (pre-treatment) and within 1 week after completion of the 3-week rTMS/sham treatment course.
  Mean change in total score on a validated autism rating scale (for example, Childhood Autism Rating Scale-2 [CARS-2]) from baseline to end of treatment, comparing active rTMS with sham in children and adolescents with autism spectrum disorder. The analysis will use mixed-effects models including fixed effects for group (active vs sham), time, and group × time interaction to estimate the treatment effect on autism symptom severity.